CLINICAL TRIAL: NCT00195351
Title: A Multicenter, Open-Label, Randomized Comparative Study of Tigecycline vs Ceftriaxone Sodium Plus Metronidazole for the Treatment of Hospitalized Subjects With Complicated Intra-abdominal Infection
Brief Title: Study Comparing Tigecycline Versus Ceftriaxone Sodium Plus Metronidazole in Complicated Intra-abdominal Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3074A1-400
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-06-10 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Appendicitis; Cholecystitis; Cross Infection; Diverticulitis; Peritonitis
Keywords: Complicated intra-abdominal infection; Appendicitis with abscess; Perforated diverticulitis; Purulent peritonitis; Complicated cholecystitis
MeSH Terms: conditions — Appendicitis; Cholecystitis; Cross Infection; Diverticulitis; Peritonitis | interventions — Tigecycline; Ceftriaxone; Metronidazole

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: tigecycline
- B (Active Comparator)
  Interventions: Drug: ceftriaxone sodium + metronidazole

INTERVENTIONS:
Drug: tigecycline — every 12 hours IV (an initial dose of 100 mg followed by 50 mg every 12 hours)
  Arms: A
Drug: ceftriaxone sodium + metronidazole — Ceftriaxone sodium 2 g once daily intravenously plus metronidazole 1 g to 2 g daily given in divided doses intravenously. Test article should be administered for a minimum of 4 days and up to 14 days at the discretion of the investigator.
  Arms: B

SUMMARY:
This is a phase 3b/4 randomized, open-label, comparative, multicenter study of the safety and efficacy of tigecycline to ceftriaxone sodium plus metronidazole in hospitalized subjects with cIAI (Complicated Intra-Abdominal Infection). Subjects with clinical signs and symptoms of cIAI will be included for enrollment. Subjects will be stratified at randomization for Acute Physiologic and Chronic Health Evaluation scale (APACHE II) score < 10 and > 10. Subjects will be followed for efficacy through the test-of-cure assessment. Safety evaluations will occur through the treatment and post-treatment periods and continue through resolution or stability of the adverse event(s).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complicated intra-abdominal infection that requires surgery within 24 hours.
* Fever over 100.4°F (38.0°C) or high white blood cell count plus other symptoms such as nausea, vomiting, abdominal pain.

Exclusion Criteria:

* Cancer
* Medicines that suppress the immune system
* Dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (57):
- United States (41):
  - Mobile, Alabama
  - Laguna Hills, California
  - Los Angeles, California
  - Orange, California
  - Palm Springs, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - West Roxbury, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Butte, Montana
  - Lincoln, Nebraska
  - Laconia, New Hampshire
  - Buffalo, New York
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Zanesville, Ohio
  - Pittsburgh, Pennsylvania
  - Corsiana, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Buenos Aires, Argentina
- Brazil (2):
  - Curitiba, Paraná
  - São Paulo, São Paulo
- Canada (10):
  - Calgary, Alberta
  - Victoria, British Columbia
  - Ajax, Ontario
  - Oshawa, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Rimouski, Quebec
  - Trois-Rivières, Quebec
- Chile (2):
  - Santiago
  - Viña del Mar
- Mexico D.F. CP, Mexico

REFERENCES:
- [Derived] Towfigh S, Pasternak J, Poirier A, Leister H, Babinchak T. A multicentre, open-label, randomized comparative study of tigecycline versus ceftriaxone sodium plus metronidazole for the treatment of hospitalized subjects with complicated intra-abdominal infections. Clin Microbiol Infect. 2010 Aug;16(8):1274-81. doi: 10.1111/j.1469-0691.2010.03122.x. PMID 20670293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited worldwide from September 2005 to February 2008.
Pre-assignment Details: Subjects were screened up to two days.
Groups:
- Tigecycline: Administered intravenously every 12 hours (an initial dose of 100 mg followed by 50 mg every 12 hours).
- Ceftriaxone Sodium + Metronidazole: Ceftriaxone sodium 2 g administered intravenously once daily plus metronidazole 1 g to 2 g daily in divided IV doses.
Period: Overall Study
Arm/Group | Tigecycline | Ceftriaxone Sodium + Metronidazole
Started | 236 | 231
Completed | 215 | 215
Not Completed | 21 | 16
Not completed — Lost to Follow-up | 9 | 9
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Protocol Deviation | 3 | 2
Not completed — Death | 3 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline | Ceftriaxone Sodium + Metronidazole | Total
Number analyzed (Participants) | 236 | 231 | 467
Age Continuous [Mean (Standard Deviation); unit: years] | 48.17 (18.05) | 48.79 (17.46) | 48.48 (17.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 72 | 165
  Male | 143 | 159 | 302
Region of Enrollment [Number; unit: participants]
  United States | 163 | 169 | 332
  Mexico | 1 | 0 | 1
  Canada | 39 | 25 | 64
  Argentina | 4 | 2 | 6
  Brazil | 23 | 23 | 46
  Chile | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Clinically Evaluable Patients With Clinical Response of Cure at Test-of-Cure (TOC) Visit.
Description: The clinical response was assigned by the investigator according to the protocol-specified guidelines. A clinical response of cure was defined as: the test article and the initial intervention (operative and/or radiologically controlled drainage procedure) resolved the intra-abdominal infection.
Time Frame: 10-21 days after the last dose of test article
Population: All patients who received ≥1 dose of study drug, who had clinical evidence of complicated intra-abdominal infection, met all inclusion and exclusion criteria, and completed TOC assessment within 8-44 days after last dose of study drug. Patients with an indeterminate assessment were excluded.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ceftriaxone Sodium + Metronidazole
Number analyzed (Participants) | 189 | 187
participants | 133 | 139
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone Sodium + Metronidazole; Test type: Superiority or Other; p = 0.009, t-test, 2 sided; Risk Difference (RD) = -4.0, 95% CI [-13.1 to 5.1]

2. Secondary Outcome: Number of Microbiologically Evaluable Patients With a Clinical Response of Cure at Test-of-Cure (TOC) Visit.
Description: as for outcome 1
Time Frame: 10-21 days after the last dose of test article
Population: All patients who received ≥1 dose, had clinical evidence of complicated intra-abdominal infection, met all inclusion/exclusion criteria, completed TOC assessment within 8-44 days after last dose, and had a baseline culture with ≥1 identified isolate that was susceptible to both study drugs. Patients with an indeterminate assessment were excluded.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ceftriaxone Sodium + Metronidazole
Number analyzed (Participants) | 138 | 137
participants | 91 | 96
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone Sodium + Metronidazole; Test type: Superiority or Other; p = 0.020, t-test, 2 sided; Risk Difference (RD) = -3.4, 95% CI [-14.5 to 7.8]

3. Secondary Outcome: Number of Patients by Microbiologic Response at Test-of-Cure (TOC) Visit.
Description: Microbiologic response assessed at patient level was combined microbiologic responses for all baseline isolates identified in intra-abdominal/blood cultures. Eradication=baseline isolate not recovered from primary infection site/blood; Presumed Eradication=no material available for culture but response was cure; Persistence=baseline isolate recovered from primary infection site/blood; Presumed Persistence=no material available for culture but response was failure; Superinfection=culture from primary infection site was positive for new isolate not identified at baseline & response was failure.
Time Frame: 10-21 days after the last dose of test article
Population: All patients who received ≥1 dose, had clinical evidence of complicated intra-abdominal infection, met all inclusion/exclusion criteria, completed TOC assessment within 8-44 days after last dose, and had baseline culture with ≥1 identified isolate that was susceptible to both study drugs. Patients with an indeterminate assessment were excluded.
Measure: Number; unit: participants
Arm/Group | Tigecycline | Ceftriaxone Sodium + Metronidazole
Number analyzed (Participants) | 138 | 137
participants
  Eradication and presumed eradication | 94 | 98
  Persistence and presumed persistence | 44 | 39
  Superinfection | 7 | 3
Statistical Analysis 1: Comparison: Tigecycline vs Ceftriaxone Sodium + Metronidazole; Test type: Superiority or Other; p = 0.015, Method of Mehrotra and Railkar; Risk Difference (RD) = -2.9, 95% CI [-13.9 to 8.1]

ADVERSE EVENTS:
Arm/Group | Tigecycline | Ceftriaxone Sodium + Metronidazole
Serious Adverse Events (participants affected / at risk) | 51 | 49
Other Adverse Events (participants affected / at risk) | 195 | 189
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tigecycline | Ceftriaxone Sodium + Metronidazole
Abscess (General disorders) | 18/236 | 13/231
Infection (General disorders) | 3/236 | 4/231
Abdominal pain (General disorders) | 3/236 | 3/231
Lymphocele (General disorders) | 0/236 | 4/231
Peritonitis (General disorders) | 1/236 | 2/231
Sepsis (General disorders) | 0/236 | 3/231
Chest pain (General disorders) | 1/236 | 1/231
Septic shock (General disorders) | 2/236 | 0/231
Hemoperitoneum (General disorders) | 0/236 | 1/231
Mesenteric fibrosis (General disorders) | 1/236 | 0/231
Retroperitoneal hemorrhage (General disorders) | 0/236 | 1/231
Traumatic hematoma (General disorders) | 1/236 | 0/231
Ileus (Gastrointestinal disorders) | 3/236 | 3/231
Intestinal obstruction (Gastrointestinal disorders) | 2/236 | 3/231
Gastrointestinal carcinoma (Gastrointestinal disorders) | 2/236 | 1/231
Cholestatic jaundice (Gastrointestinal disorders) | 2/236 | 0/231
Constipation (Gastrointestinal disorders) | 0/236 | 1/231
Diarrhea (Gastrointestinal disorders) | 1/236 | 0/231
Gastrointestinal disorder (Gastrointestinal disorders) | 0/236 | 1/231
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1/236 | 0/231
Hematemesis (Gastrointestinal disorders) | 0/236 | 1/231
Intestinal necrosis (Gastrointestinal disorders) | 1/236 | 0/231
Melena (Gastrointestinal disorders) | 0/236 | 1/231
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2/236 | 5/231
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/236 | 3/231
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1/236 | 1/231
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0/236 | 2/231
Carcinoma of the lung (Respiratory, thoracic and mediastinal disorders) | 1/236 | 0/231
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/236 | 1/231
Pulmonary embolus (Cardiac disorders) | 3/236 | 1/231
Atrial fibrillation (Cardiac disorders) | 2/236 | 0/231
Deep vein thrombosis (Vascular disorders) | 2/236 | 0/231
Hypotension (Cardiac disorders) | 1/236 | 1/231
Myocardial infarct (Cardiac disorders) | 0/236 | 2/231
Cerebral ischemia (Vascular disorders) | 1/236 | 0/231
Cerebrovascular accident (Vascular disorders) | 1/236 | 0/231
Congestive heart failure (Cardiac disorders) | 0/236 | 1/231
Coronary artery disorder (Cardiac disorders) | 0/236 | 1/231
Heart arrest (Cardiac disorders) | 1/236 | 0/231
Hemorrhage (Vascular disorders) | 1/236 | 0/231
Mesenteric venous occousion (Vascular disorders) | 1/236 | 0/231
Healing abdominal (Metabolism and nutrition disorders) | 3/236 | 1/231
Acidosis (Metabolism and nutrition disorders) | 0/236 | 1/231
Blood urea nitrogen increased (Metabolism and nutrition disorders) | 0/236 | 1/231
Thrombocythemia (Blood and lymphatic system disorders) | 2/236 | 0/231
Anemia (Blood and lymphatic system disorders) | 0/236 | 1/231
International normalized ratio increased (Blood and lymphatic system disorders) | 1/236 | 0/231
Acute kidney failure (Renal and urinary disorders) | 0/236 | 1/231
Pyelonephritis (Renal and urinary disorders) | 1/236 | 0/231
Urinary retention (Renal and urinary disorders) | 1/236 | 0/231
Trauma (General disorders) | 0/236 | 1/231
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Tigecycline | Ceftriaxone Sodium + Metronidazole
Nausea (Gastrointestinal disorders) | 91/236 | 64/231
Vomiting (Gastrointestinal disorders) | 55/236 | 41/231
Diarrhea (Gastrointestinal disorders) | 42/236 | 40/231
Constipation (Gastrointestinal disorders) | 14/236 | 14/231
Ileus (Gastrointestinal disorders) | 8/236 | 16/231
Abdominal distension (Gastrointestinal disorders) | 5/236 | 11/231
Dyspepsia (Gastrointestinal disorders) | 9/236 | 4/231
Oral moniliasis (Gastrointestinal disorders) | 8/236 | 1/231
Abdominal pain (General disorders) | 22/236 | 16/231
Abscess (General disorders) | 23/236 | 15/231
Headache (General disorders) | 14/236 | 22/231
Fever (General disorders) | 17/236 | 18/231
Infection (General disorders) | 17/236 | 9/231
Generalized edema (General disorders) | 1/236 | 7/231
Hypokalemia (Metabolism and nutrition disorders) | 16/236 | 21/231
Healing abdominal (Metabolism and nutrition disorders) | 9/236 | 8/231
Hyperglycemia (Metabolism and nutrition disorders) | 9/236 | 8/231
Peripheral edema (Metabolism and nutrition disorders) | 9/236 | 7/231
Hypoproteinemia (Metabolism and nutrition disorders) | 11/236 | 4/231
Amylase increased (Metabolism and nutrition disorders) | 8/236 | 4/231
Hypophophatemia (Metabolism and nutrition disorders) | 3/236 | 9/231
SGPT increased (Metabolism and nutrition disorders) | 7/236 | 5/231
Insomina (Nervous system disorders) | 23/236 | 24/231
Anxiety (Nervous system disorders) | 7/236 | 12/231
Confusion (Nervous system disorders) | 8/236 | 2/231
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 9/236 | 8/231
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6/236 | 10/231
Pulmonary physical findings (Respiratory, thoracic and mediastinal disorders) | 7/236 | 6/231
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5/236 | 7/231
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4/236 | 7/231
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0/236 | 7/231
Thrombocythemia (Blood and lymphatic system disorders) | 13/236 | 15/231
Anemia (Blood and lymphatic system disorders) | 16/236 | 8/231
Leukocytosis (Blood and lymphatic system disorders) | 19/236 | 4/231
Hypertension (Cardiac disorders) | 9/236 | 11/231
Deep vein thrombosis (Vascular disorders) | 8/236 | 1/231
Pruritus (Skin and subcutaneous tissue disorders) | 13/236 | 12/231
Rash (Skin and subcutaneous tissue disorders) | 4/236 | 7/231
Local reaction to procedure (Surgical and medical procedures) | 18/236 | 14/231
Taste perversion (General disorders) | 2/236 | 9/231

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.